CLINICAL TRIAL: NCT04001933
Title: CenteringPregnancy Oral Health Promotion (CPOP) Clinical Trial
Brief Title: CenteringPregnancy Oral Health Promotion
Acronym: CPOP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The onset of COVID-19 shut down San Francisco in March 2020, resulting in immediate suspension of group prenatal care at our clinic sites. This continued suspension prevented the conduct of study activities, which resulted in study termination.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-029-E; 1U01DE027340-01 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-28 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Oral Health
Keywords: Pregnancy; Oral Health; Maternal Oral Health; Infant Oral Health

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): CPOP Intervention (see below).
  Interventions: Other: CPOP Intervention
- Control Arm (No Intervention): Usual care.

INTERVENTIONS:
Other: CPOP Intervention — The intervention consists of two 15-minute interactive modules (maternal and infant OH), integrated into 2 group prenatal care sessions. Led by trained prenatal care providers (facilitators), the maternal module includes discussion of common OH problems during pregnancy, importance of OH, importance and safety of OH care during pregnancy, hands-on skills-building activities of learning and practicing proper tooth brushing and self-assessment of gum health, and presentation of illustrated flossing and OH promotion guides. The infant module includes discussion of infant oral hygiene, avoiding saliva sharing, proper nutrition, and importance of a dental visit by the first birthday. Activities in both modules utilize separate tool kits including tooth brushes, fluoride toothpaste, and other supplies.
  Arms: Intervention Arm

SUMMARY:
A five-year, Phase III, multi-site, cluster randomized controlled clinical trial will evaluate the efficacy of the CenteringPregnancy (CP) Oral Health Promotion (CPOP) intervention. Intervention and control groups will be drawn from 6 CP sites. Prenatal care facilitators will conduct the intervention in group prenatal care sessions. With an average of 4 CP facilitators per site (24 facilitators), conducting 2-3 CP groups each (48-72 CP groups with 8 mother/child dyads per group), the total study population will be approximately 384 dyads. CP facilitators will be randomly assigned to either the: 1) intervention arm and deliver the CPOP intervention; or 2) control arm and deliver the usual CP curriculum. The CPOP intervention consists of two 15-minute modules: 1) maternal oral health (OH) and 2) infant OH. The data collection will continue through 12 months postpartum. For the maternal OH module, pre- and post-intervention dental exams of gingival OH and Plaque Levels, and knowledge, attitudes and behavior (KAB) questionnaires during the prenatal period will be used to assess maternal OH outcomes. For the infant OH module, pre and post-module KAB questionnaires will be completed during the prenatal period. Infant OH risk status - the presence of caries-causing bacteria (mutans streptococci and Lactobacilli) in saliva of both mother and infant will be assessed when the infant is 12 months of age to determine differences in study arms.

ELIGIBILITY:
Inclusion Criteria:

Women:

* speak, read, or write in English or Spanish
* enrolled in CP prenatal group care identified as study group
* free of any condition that requires them to take antibiotic or antibacterial medication prior to dental procedures
* provide informed consent

Babies:

* healthy with no acute or chronic medical conditions, especially those conditions that may have resulted in hospitalizations and subsequent exposure to pathologic microorganisms
* free of any condition requiring antibiotic treatment currently or within the past three months.
* mothers provide informed consent for their children at baseline

Exclusion Criteria:

- none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in percent of periodontal probing sites that bleed upon probing | 12 weeks follow-up
  Based on clinical dental exams conducted before the maternal oral health module and approximately 12 weeks following the maternal module, comparisons between the Intervention and Control groups will be conducted to determine differences in change in the percent of periodontal probing sites that bleed upon probing.
Change in percent of periodontal probing sites that probe at ≥4mm depth | 12 weeks follow-up
  Based on clinical dental exams conducted before the maternal oral health module and approximately 12 weeks following the maternal module, comparisons between the Intervention and Control groups will be conducted to determine differences in change in the percent of periodontal probing sites that probe at ≥4mm depth.
Change in plaque levels at 24 sites | 12 weeks follow-up
  Based on clinical dental exams conducted before the maternal oral health module and approximately 12 weeks following the maternal module, comparisons between the Intervention and Control groups will be conducted to determine differences in change in plaque levels at 24 sites (4 sites on 6 teeth) using the Plaque Index. Each site is scored from 0-3 (0=no plaque; 3=heavy plaque), yielding a score between 0 and 72.
Incidence of salivary Mutans Streptococci in infants at 12 months of age | 1-year follow-up postpartum
  Based on results of assays of infant saliva specimens collected at 12 months of age, comparisons between infants whose mothers were in the Intervention versus the Control groups will be conducted to determine differences in the incidence of Mutans Streptococci.

SECONDARY OUTCOMES:
Change in maternal oral health knowledge | 12 week follow-up
  Self reported oral health knowledge questionnaire which includes 12 dichotomous items (0-1) for a total between 0 and 12 used for comparisons between the Intervention and Control groups.
Change in maternal oral health attitude | 12 week follow-up
  Self reported oral health attitude questionnaire which includes 8 items scored 1-4 (1=Not at all important; 4=Very important) for a total between 8 and 32 used for comparisons between the Intervention and Control groups.
Change in maternal oral health behavior | 12 week follow-up
  Self reported oral health behavior questionnaire which includes 4 items scored as either correct or incorrect (0=Incorrect; 1=Correct) for a total between 0-4 used for comparisons between the Intervention and Control groups.
Change in maternal knowledge regarding infant oral health | 2 week follow-up
  Self reported infant oral health knowledge questionnaire which includes 10 dichotomous items (0-1) for a total between 0 and 10 used for comparisons between the Intervention and Control groups.
Change in maternal attitude regarding infant oral health | 2 week follow-up
  Self reported infant oral health attitude questionnaire which includes 8 items scored 1-4 (1=Not at all important; 4=Very important) for a total between 8 and 32 used for comparisons between the Intervention and Control groups.
Incidence of salivary Lactobacillus in infants at 12 months of age | 1 year follow-up postpartum
  Based on results of assays of infant saliva specimens collected at 12 months of age, comparisons between infants whose mothers were in the Intervention versus the Control groups will be conducted to determine differences in the incidence of Lactobacillus.
Mediation outcomes for maternal oral health are maternal oral health knowledge | 12 week follow-up
  Evaluation of maternal oral health knowledge as a mediator of the association between treatment arm and plaque, probing and bleeding.
Mediation outcomes for maternal oral health are maternal oral health attitudes (importance and self-efficacy) | 12 week follow-up
  Evaluation of maternal oral health attitudes as a mediator of the association between treatment arm and plaque, probing and bleeding.
Mediation outcomes for maternal oral health are maternal oral health behaviors (ADA-recommended tooth brushing practices and flossing) | 12 week follow-up
  Evaluation of maternal oral health behaviors as a mediator of the association between treatment arm and plaque, probing and bleeding.
Mediation outcomes for infant oral health risk are infant oral health-related knowledge | 1 year follow-up postpartum
  Evaluation of maternal knowledge of infant oral health as a mediator of the association between treatment arm and infant MS and LB.
Mediation outcomes for infant oral health risk are infant oral health-related attitudes (importance and self-efficacy) | 1 year follow-up postpartum
  Evaluation of maternal attitudes toward infant oral health as a mediator of the association between treatment arm and infant MS and LB.
Mediation outcomes for infant oral health risk are infant oral health-related behaviors (importance and self-efficacy) | 1 year follow-up postpartum
  Evaluation of maternal behaviors toward infant oral health as a mediator of the association between treatment arm and infant MS and LB.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Berens, DDS, MPH, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04001933/Prot_SAP_001.pdf